CLINICAL TRIAL: NCT05584800
Title: A Phase I/II Dose Escalation, Tolerability, Safety, Pharmacokinetics and Multiple Cohort Expansion Study of ZGGS18 in Patients With Advanced Solid Tumors
Brief Title: Study of ZGGS18 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZGGS18-001
Record Dates: First submitted 2022-10-10; First posted 2022-10-18 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental)
  Interventions: Biological: ZGGS18 for Injection
- Dose Expansion (Experimental): Tumor type: colorectal cancer，pancreatic cancer
  Interventions: Biological: ZGGS18 for Injection

INTERVENTIONS:
Biological: ZGGS18 for Injection — 0.3 mg/kg, 1 mg/kg, 3 mg/kg, 6 mg/kg, 10 mg/kg, 15 mg/kg and 20 mg/kgof ZGGS18，intravenous infusion, once every 2 weeks.
  Arms: Dose Escalation
Biological: ZGGS18 for Injection — Recommended Phase 2 Dose (RP2D) (to be determined) of ZGGS18，intravenous infusion, once every 2 weeks.
  Arms: Dose Expansion

SUMMARY:
A clinical study to assess dose escalation, tolerance, safety, pharmacokinetics, and multi cohort expansion of ZGGS18 in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced solid tumors, who had failed the available standard treatments or no standard treatment or intolerance to standard treatment;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
* Life expectancy ≥ 3 months;
* Must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors 1.1(RECIST1.1). For lesions that have received radiation therapy, only after the progression of the lesions, they can be considered measurable lesions.

Exclusion Criteria:

* The investigator considers that any subjects are not suitable to participate in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Tolerability of ZGGS18 | 28 days
  Dose limiting toxicity, number of participants with abnormal laboratory values and/or adverse events that are related to treatment
Safety of ZGGS18 | Through study completion, an expected average of 3 years
  Number of participants with adverse events/abnormal laboratory values that are related to treatment

SECONDARY OUTCOMES:
Pharmacokinetic characteristics of ZGGS18 | Through Phase I study completion, an expected average of 1 year
  Peak Plasma Concentration (Cmax)
Pharmacokinetic characteristics of ZGGS18 | Through Phase I study completion, an expected average of 1 year
  Time to maximum concentration (Tmax)
Pharmacokinetic characteristics of ZGGS18 | Through Phase I study completion, an expected average of 1 year
  Clearance (CL/F)
Pharmacokinetic characteristics of ZGGS18 | Through Phase I study completion, an expected average of 1 year
  Area under drug concentration-time curve
Pharmacokinetic characteristics of ZGGS18 | Through Phase I study completion, an expected average of 1 year
  Elimination rate constant (Ke)
Pharmacokinetic characteristics of ZGGS18 | Through Phase I study completion, an expected average of 1 year
  Elimination half-life (t1/2)
Immunogenicity of ZGGS18 | Through study completion, an expected average of 3 years
  Detection of anti-drug antibodies, if positive, further detection of neutralizing antibodies. Counting the number of patients and incidence of anti-drug antibodies and neutralizing antibodies
Efficacy of ZGGS18 | Through study completion, an expected average of 3 years
  Objective response rate
Efficacy of ZGGS18 | Through study completion, an expected average of 3 years
  Progression-free survival
Efficacy of ZGGS18 | Through study completion, an expected average of 3 years
  Disease control rate
Efficacy of ZGGS18 | Through study completion, an expected average of 3 years
  Duration of response
Efficacy of ZGGS18 | Through study completion, an expected average of 3 years
  Time to response
Efficacy of ZGGS18 | Through study completion, an expected average of 3 years
  Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Director — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No